CLINICAL TRIAL: NCT06856083
Title: Development of Innovative Strategies for Improving Life Satisfaction in Elderly With Suicidal Ideation: The Impact of Gamified VR Sports Training
Brief Title: Gamified VR Sports for Elderly Suicidal Ideation
Acronym: VR-LIFE-SI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Zinat Ebrahimi, Assistant Professor, Department of Physical Education and Sport Science, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VR-LIFE-SI-2025
Record Dates: First submitted 2025-02-11; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Suicidal Ideation; Depression; Mental Health Issue
Keywords: Gamified virtual reality exercises; Elderly mental health; Suicidal thoughts intervention; Physical activity in older adults; VR sports training; Depression reduction; Life expectancy improvement; Quasi-experimental study; Non-pharmacological intervention; Interactive exercise program; Mental health support for seniors; Gamification in healthcare; Elderly population study; Community engagement through exercise; Innovative health interventions
MeSH Terms: conditions — Suicidal Ideation; Depression | interventions — Aging; Mental Health

STUDY DESIGN:
Intervention Model Description: This study employs a quasi-experimental interventional model designed to evaluate the impact of gamified virtual reality sports exercises on mental health and life expectancy in elderly individuals (aged 60 and over) experiencing suicidal thoughts. Participants will be randomly assigned to either the experimental group, which will engage in VR-based sports training sessions utilizing gamification elements, or the control group, which will participate in conventional sports exercises without immersive technology or gamification.
  The intervention aims to enhance physical activity engagement through an interactive and supportive environment, fostering community and social interaction among participants. Data will be gathered through baseline assessments and follow-up evaluations to gauge changes in mental health indicators, including suicidal ideation and perceived life expectancy.
Who Masked: Participant, Care Provider
Masking Description: In this study, participants will not be fully masked to group assignment due to the nature of the intervention. However, to mitigate bias in reporting and assessment, care providers who conduct the outcome assessments will be masked to the group assignments of the participants. This means that the assessors evaluating participants' mental health and life expectancy outcomes will not know whether individuals belong to the experimental group (engaging in VR-based sports exercises) or the control group (participating in traditional exercises).
  Additionally, researchers conducting the data analysis will also remain blinded to group allocations to ensure objective evaluation of results and reduce any potential biases during interpretation. This masking approach is designed to preserve the integrity of the study findings and ensure that the effects of the intervention are accurately attributed to the gamified VR sports exercises.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamified Virtual Reality Sports Exercise Program for Elderly Individuals with Suicidal Thoughts (Experimental): Participants will engage in a gamified virtual reality (VR) sports exercise program specifically designed for elderly individuals experiencing suicidal thoughts. The intervention consists of structured, immersive VR sessions that incorporate various sports activities tailored to accommodate the physical abilities of the participants. These sessions will utilize gamification elements, including points, rewards, and friendly competition, to enhance motivation and engagement.
  Participants will join weekly VR exercise sessions guided by trained facilitators who will provide support and encouragement throughout the program. The aim is to foster social interaction among participants, creating a sense of community and reducing feelings of loneliness. Each session will last approximately 60 minutes and will include warm-up exercises, the main VR activity, and a cooldown
  Interventions: Behavioral: Traditional Sports Exercise Program for Elderly Individuals with Suicidal Thoughts
- Active Comparator: Traditional Sports Exercise Program for Elderly Individuals with Suicidal Thought (Experimental): Participants will engage in a traditional sports exercise program aimed at elderly individuals experiencing suicidal thoughts. The intervention consists of structured physical activity sessions that include a variety of low-impact sports and exercises designed for older adults. These activities will be conducted in a supportive group setting to foster social interaction and community engagement.
  The sessions will be led by experienced facilitators who specialize in elderly fitness and mental health. Each session will last approximately 60 minutes and will include a warm-up, the main exercise component, and a cooldown period to promote physical well-being and relaxation. Participants will be encouraged to engage at their own pace, ensuring that individual capabilities and comfort levels are respected.
  Behavioral: Traditional Sports Exercise Program Structured physical activity sessions led by experienced facilitators. Low-impact sports and exercises tailored for older adults.
  Interventions: Behavioral: Gamified Virtual Reality Sports Exercise Program

INTERVENTIONS:
Behavioral: Gamified Virtual Reality Sports Exercise Program — Participants in the experimental group will participate in a variety of sports exercises designed in a virtual reality environment utilizing gamification elements to enhance engagement. The intervention will include:
  * Structured virtual reality sports sessions guided by specially trained facilitators.
  * Use of gamified features such as rewards, points, and friendly competition to stimulate motivation.
  * Incorporation of social elements where participants can interact with each other during sessions to foster community and support.
  Other Names: VR-Based Gamified Exercise Program; Immersive VR Sports Training for Elderly; Virtual Reality Gamification for Mental Health
  Arms: Active Comparator: Traditional Sports Exercise Program for Elderly Individuals with Suicidal Thought
Behavioral: Traditional Sports Exercise Program for Elderly Individuals with Suicidal Thoughts — participants will engage in a traditional sports exercise program aimed at elderly individuals experiencing suicidal thoughts. The intervention consists of structured physical activity sessions that include a variety of low-impact sports and exercises designed for older adults. These activities will be conducted in a supportive group setting to foster social interaction and community engagement.
  The sessions will be led by experienced facilitators who specialize in elderly fitness and mental health. Each session will last approximately 60 minutes and will include a warm-up, the main exercise component, and a cooldown period to promote physical well-being and relaxation. Participants will be encouraged to engage at their own pace, ensuring that individual capabilities and comfort levels are respected.
  Other Names: Conventional Physical Activity Program; Low-Impact Sports for Elderly; Group-Based Exercise for Mental Health
  Arms: Gamified Virtual Reality Sports Exercise Program for Elderly Individuals with Suicidal Thoughts

SUMMARY:
Detailed Description:

This quasi-experimental study investigates the effectiveness of a gamified sports exercise intervention delivered through virtual reality (VR) to improve mental health and life expectancy in elderly individuals aged 60 and over who are experiencing suicidal thoughts. The study aims to address the following research questions:

How do gamified sports exercises in a virtual reality environment impact the mental health of elderly individuals with suicidal thoughts? What differences in mental health outcomes are observed between participants engaging in gamified VR exercises and those participating in conventional sports exercises?

The study design involves two groups:

Experimental Group: Participants will engage in VR-based sports training sessions that incorporate gamification elements, such as rewards, competition, and interactive challenges.

Control Group: Participants will participate in traditional sports exercises without gamification or VR components.

Procedures:

Baseline Assessment: All participants will complete a life expectancy questionnaire and standardized mental health assessments to establish baseline data.

Intervention:

The experimental group will undergo a series of VR-based sports training sessions, designed to be engaging and immersive, with gamified elements to enhance motivation and adherence.

The control group will participate in conventional sports exercises, such as light aerobic activities or stretching, delivered in a standard, non-gamified format.

Post-Intervention Assessment: Mental health outcomes, including changes in suicidal ideation, life satisfaction, and overall well-being, will be evaluated using validated questionnaires and scales.

Expected Outcomes:

The study hypothesizes that the experimental group will demonstrate significant improvements in mental health outcomes, including reduced suicidal ideation and increased life satisfaction, compared to the control group. The findings aim to provide evidence-based insights into the potential of gamified VR interventions as a non-pharmacological strategy to enhance the well-being of elderly individuals at risk for suicide.

This study contributes to the growing body of research on innovative approaches to mental health support for vulnerable populations, with a focus on leveraging technology to improve quality of life and reduce suicide risk among the elderly.

DETAILED DESCRIPTION:
Detailed Description

Background Aging is associated with an increased incidence of chronic diseases and mental health issues, including depression and suicidal ideation. Elderly individuals (aged 60 and over) represent a vulnerable population at heightened risk for suicide. Research indicates that physical activity plays a crucial role in improving both mental and physical health outcomes. However, many elderly individuals encounter significant barriers to regular participation in physical exercises, such as low motivation and limited access to facilities.

Emerging technologies, such as gamification and virtual reality (VR), have shown promise in enhancing engagement in health-related behaviors. Gamification-integrating game-like elements into non-game contexts-has been recognized as a potent tool to motivate individuals to participate in physical activities. VR offers an immersive experience that may further enhance the appeal of physical exercises for older adults.

Purpose This study aims to evaluate the effectiveness of a gamified sports exercise program in a virtual reality environment as a means to improve mental health and life satisfaction among elderly individuals experiencing suicidal ideation. The intervention seeks to create an engaging and supportive environment to reduce suicidal ideation and increase overall life satisfaction within this demographic.

Study Design This is a quasi-experimental study with pre-test and post-test assessments. Participants will be randomly assigned to either an experimental group that engages in VR-based sports exercises or a control group that participates in conventional sports activities without gamified elements.

Intervention

Participants in the experimental group will engage in sports exercises designed in a virtual reality environment, incorporating gamification elements to enhance engagement. The intervention includes:

Structured virtual reality sports sessions guided by trained facilitators.

Gamified features such as rewards, points, and friendly competition to stimulate motivation.

Social interaction elements where participants can engage with each other during sessions to foster community and support.

The control group will participate in traditional physical activity sessions without VR or gamification.

Assessments

Baseline assessments will be conducted before the interventions, with follow-up assessments after the 8-week intervention period. The following tools will be utilized:

Life Expectancy Questionnaire: A validated tool to assess participants' perceptions of their future and overall well-being.

Suicidal Ideation Scale: A standard scale to measure the severity of suicidal thoughts.

Depression Inventory: To assess levels of depressive symptoms before and after the intervention.

Data Analysis Data will be analyzed using appropriate statistical methods to assess the effectiveness of the gamified sports exercise program compared to conventional exercises. Primary outcomes will focus on changes in mental health indicators, including suicidal ideation, life expectancy perceptions, and overall quality of life.

Expected Outcomes

The study anticipates that participation in the gamified virtual reality sports exercises will lead to:

A significant reduction in suicidal thoughts and depressive symptoms among participants.

Improved perceptions of life expectancy among elderly individuals.

Higher rates of physical activity engagement in the experimental group compared to the control group.

Significance The findings of this study are expected to contribute valuable knowledge to the field of elderly mental health, particularly for strategies aimed at reducing suicide risks. By addressing the interplay of mental health and physical activity, the research aims to provide evidence for innovative intervention strategies that can enhance the quality of life for vulnerable elderly populations.

Ethical Considerations The study will adhere to ethical guidelines for research. Informed consent will be obtained from all participants (or their guardians) before enrollment, ensuring they fully understand the study's purpose, procedures, and their right to withdraw at any time.

Key Changes:

Removed Duplicate Information:

Removed eligibility criteria and sample size details, as these are recorded in other data elements.

Focused on providing extended technical details about the intervention, assessments, and data analysis.

Technical and Extended Description:

Added more technical details about the VR-based sports exercises, gamification elements, and assessment tools.

Ensured the description aligns with the protocol's purpose and design without repeating information from other sections.

Improved Flow and Readability:

Organized content into clear sections for better readability and alignment with protocol requirements.

ELIGIBILITY:
Inclusion Criteria:

* Elderly men aged 60 years and older
* Suicidal thoughts confirmed by psychological evaluation
* Symptoms of depression and loneliness
* Informed consent provided by participant or family
* Residency in Tehran, Iran

Exclusion Criteria:

* Severe cognitive impairment or dementia
* Current therapeutic interventions for suicidal ideation or mental health issues
* Acute medical conditions requiring immediate attention
* History of severe substance abuse or dependence
* Significant physical disabilities preventing basic physical activity

Min Age: 58 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2023-10-14 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Suicidal Ideation as Measured by the Beck Scale for Suicide Ideation (BSSI) | Baseline and post-intervention (2 months).
  Description: The Beck Scale for Suicide Ideation (BSSI) is a validated 21-item questionnaire used to assess the intensity and frequency of suicidal thoughts. Scores range from 0 to 38, with higher scores indicating greater severity of suicidal ideation. This measure will be administered at baseline and after 2 months of participation to evaluate changes in suicidal ideation among elderly participants.
Change in Depressive Symptoms as Measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline and post-intervention (2 months).
  Description: The Patient Health Questionnaire-9 (PHQ-9) is a validated 9-item questionnaire used to assess the severity of depressive symptoms based on DSM-5 criteria. Scores range from 0 to 27, with higher scores indicating more severe depression. This measure will be administered at baseline and after 2 months of participation to evaluate changes in depressive symptoms among elderly participants.

CONTACTS AND LOCATIONS:
Overall Officials: Zinat Dr Zinat Ebrahimi, Professor, Principal Investigator — Islamic Azad University
Locations (1):
- Department of Physical Education and Sport Science, Faculty of Humanities and Literature, Sanandaj Branch, Islamic Azad University, Sanandaj, Iran., Sanandaj, Kurdistan Province, Iran

IPD SHARING:
Plan to Share IPD: No
Due to persistent technical difficulties in providing a functional web address for the IPD sharing plan on the clinical trial site, interested parties are encouraged to contact zin368@gmail.com for further information. We have encountered issues that prevent the proper display or access of the sharing link, necessitating this alternative means of communication.

REFERENCES:
- [Background] Chambers, L.W. and L.W. Chambers, Prevalence and monetary costs of dementia in Canada. 2016: Miscellaneous Agency.